CLINICAL TRIAL: NCT04160195
Title: T Cells Expressing Fully-human Anti-CD19 and Anti-CD20 Chimeric Antigen Receptors for Treating B-cell Malignancies and Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The original principal investigator left the National Institutes of Health (NCI) and the decision was made to close the study to enrollment.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Kochenderfer, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200008; 20-C-0008
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Non-hodgkins; Chronic Lymphocytic Leukemia; B-Cell Chronic Lymphocytic Leukemia
Keywords: Autologous T Cells Infusion; Hu1928-Hu20BB; Hodgkin Reed-Sternberg Cells; Adoptive T Cell Therapy; Gene Therapy
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Automobiles; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Conditioning chemotherapy plus Chimeric Antigen Receptors (CAR) T-cells dose escalation (Active Comparator): All participants will be receiving escalating dose of Anti-cluster of differentiation 19 (CD19) and anti-cluster of differentiation 20 (CD20) CAR T cells/kg + conditioning chemotherapy
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptors (CAR) and Anti-cluster of differentiation 20 (CD20)-CAR T cells; Drug: Cyclophosphamide; Drug: Fludarabine
- 2/Conditioning chemotherapy plus Chimeric Antigen Receptors (CAR) T-cells expansion phase (Active Comparator): Maximum tolerated dose (MTD) dose of Anti-cluster of differentiation 19 (CD19) and anti-cluster of differentiation 20 (CD20) CAR T cells/kg + Conditioning chemotherapy
  Interventions: Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptors (CAR) and Anti-cluster of differentiation 20 (CD20)-CAR T cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptors (CAR) and Anti-cluster of differentiation 20 (CD20)-CAR T cells — Dose-escalation trial starting dose: 0.66 x10^6 CAR+ T cells/kg (weight-based dosing one time) (up to a maximum dose of 10x10^6 CAR+ T cells/kg based on cohort) infuse on day 0
Drug: Cyclophosphamide — 500 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3
  Other Names: Cytoxan
Drug: Fludarabine — 30 mg/m^2 intravenous (IV) infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
  Other Names: Fludara

SUMMARY:
Background:

-Cluster of differentiation 19 (CD19) and cluster of differentiation 20 (CD20) are often found on certain cancer cells. Researchers think that a person's T cells can be modified in a lab to kill cells that have CD19 and CD20 on the surface.

Objective:

-To see if it is safe to give anti-CD19 and anti-CD20 CAR T cells to people with a B cell cancer or Hodgkin lymphoma.

Eligibility:

-People ages 18 and older with a B cell cancer or Hodgkin lymphoma that has not been controlled with standard therapies

Design:

* Participants will be screened under protocol 01C0129 with:
* Medical history
* Physical exam
* Blood and heart tests
* Bone marrow biopsy: A needle is inserted into the participant's hip bone to remove a small amount of marrow.

Scans

* Participants will have apheresis: Blood will be removed through a vein. The blood with circulate through a machine that removes the T cells. The rest of the blood will be returned to the participant.
* Once a day for 3 days before they get the T cells, participants will receive chemotherapy through a vein.
* Participants will receive the T cells through a vein. They will stay in the hospital for at least 9 days.
* Participants may have a lumbar puncture: A needle will remove fluid from the spinal cord.
* Participants may have a tumor biopsy.
* Participants will repeat the screening tests throughout the study.
* Participants will have follow-up visits 2 weeks after infusion; monthly for 4 months; at 6, 9, and 12 months; every 6 months for 3 years; and then annually for 5 years. Participants will then be contacted annually for 15 years.

DETAILED DESCRIPTION:
Background:

* Improved treatments for a variety of treatment-resistant malignancies including B-cell lymphomas, and chronic lymphocytic leukemia (CLL) and Hodgkin lymphoma are needed.
* A particular need is development of new treatments for chemotherapy-refractory B-cell malignancies.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T cells genetically modified to express CARs targeting the B-cell antigen CD19 have caused complete remissions in patients with leukemia or lymphoma. These results have established anti-cluster of differentiation 19 (CD19) CAR T cells as an important therapy for relapsed lymphoma, but only about 40% of patients receiving anti-CD19 CAR T cells have durable complete remissions.
* Most B-cell malignancies express CD19 and cluster of differentiation 20 (CD20), but expression of CD19 and CD20 can be lost or diminished.
* The malignant cells of Hodgkin lymphoma, Hodgkin Reed-Sternberg cells, originate from B cells, which is the rationale for treating Hodgkin lymphoma with T cells targeting CD19 and CD20.
* CD19 and CD20 are not expressed by normal cells except for B cells and some plasma cells.
* We have constructed a novel gene therapy construct that encodes a fully-human anti-CD19 CAR with a cluster of differentiation 28 (CD28) domain and a fully-human anti-CD20 CAR with a 4-1BB (cluster of differentiation 37) domain.
* T cells expressing this CAR construct, called Hu1928-Hu20BB, can specifically recognize CD19 and CD20-expressing target cells in vitro and eradicate CD19 or CD20-expressing tumors in mice.
* One CAR expressed in this CAR construct, Hu19-CD828Z has been tested in humans before. The other CAR in the total construct, Hu20-CD8BBZ, has not been tested in humans before.
* Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of normal B cells is probable, and unknown toxicities are also possible.

Objectives:

Primary

-Determine the safety and feasibility of administering T cells expressing a novel fully-human anti- CD19 and anti-CD20 CAR construct to patients with advanced B-cell malignancies and Hodgkin lymphoma.

Exploratory

* Evaluate serum cytokine levels and associations with anti-malignancy efficacy and toxicity
* Evaluate clinical predictors of anti-lymphoma responses and toxicity.
* Evaluate phenotype of infused CAR T cells and CAR T cells from the blood of patients.

Eligibility:

* Patients must have any B-cell lymphoma, or CLL/small lymphocytic lymphoma (SLL), Gray-zone lymphoma, nodular lymphocyte-predominance Hodgkin lymphoma, or classical Hodgkin lymphoma with any CD19 or CD20 expression on Reed-Sternberg cells. Lower grade lymphomas transformed to diffuse large B-cell lymphoma (DLBCL) are potentially eligible as is primary mediastinal B-cell lymphoma and all other subtypes of DLBCL. Burkitt and mantle cell lymphoma are potentially eligible.
* Patients must have malignancy that is measurable on a computed tomography (CT) scan or by flow cytometry of bone marrow or blood.
* Patients must have a creatinine of 1.5 mg/dL or less and a normal cardiac ejection fraction.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 is required.
* No active infections are allowed including hepatitis B or hepatitis C.
* Absolute neutrophil count>=1000/mL, platelet count>=50,000/mL, hemoglobin>=8g/dL
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and protocol-required leukapheresis or CAR T-cell infusion. Thirty days must elapse from therapy with antibodies targeting CD19 or CD20 and CAR T-cell infusion.
* The patient's malignancy will need to be assessed for CD19 and C20 expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). If unstained, paraffin-embedded bone marrow or lymphoma tissue sections are available from prior biopsies, these can be used to determine CD19 and CD20 expression by immunohistochemistry; otherwise, patients will need to come to the NIH for a biopsy to determine CD19 and CD20 expression. The sample for CD19 and CD20 expression must come from a biopsy obtained after any CD19 or CD20-targeted therapies such as monoclonal antibodies if such antibodies or CAR T-cell therapies have been received by the patient.
* For classical Hodgkin lymphoma only, a biopsy from any time from any institution that shows any CD19 or CD20 expression on Reed-Sternberg cells is adequate for eligibility. CD19 or CD20 expression on the Reed-Sternberg cells that is weak or only present on some Reed-Sternberg cells by immunohistochemistry is compatible with protocol eligibility.
* For all lymphoma types except for classical Hodgkin lymphoma, either CD19 or CD20 expression must be uniform. Uniform CD19 or CD20 expression is defined as no obvious lymphoma population lacking antigen expression can be present. Antigen expression can be assessed by either immunohistochemistry or flow cytometry.

Design:

* This is a phase I dose-escalation trial
* Patients will undergo leukapheresis
* T-cells obtained by leukapheresis will be genetically modified to express the Hu1928-Hu20BB CAR construct.
* Patients will receive a lymphocyte-depleting chemotherapy conditioning regimen with the intent of enhancing the activity of the infused CAR-expressing T cells.
* The chemotherapy conditioning regimen is cyclophosphamide 500 mg/m squared daily for 3 days and fludarabine 30 mg/m squared daily for 3 days. Fludarabine will be given on the same days as the cyclophosphamide.
* Two days after the chemotherapy ends, patients will receive an infusion of anti-CAR-expressing T cells.
* The initial dose level of this dose-escalation trial will be 0.66x10^6 CAR+ T cells/kg of recipient bodyweight.
* The cell dose administered will be escalated until a maximum tolerated dose is determined.
* Following the T-cell infusion, there is a mandatory 9-day inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks, 16 days (neurologic checks), 21 days (neurologic checks) and 1, 2, 3, 4, 6, 9, and 12 months after the CAR T- cell infusion; less frequent follow-up is required more than 1 year after infusion. Long-term gene-therapy follow-up for a total of 15 years after infusion is required.

ELIGIBILITY:
* INCLUSION CRITERIA:

MALIGNANCY CRITERIA:

Note: As of approval of Amendment A, no patients with Hodgkin lymphoma can be enrolled until at least 6 patients with B-cell malignancies are treated without incidence of Guillain-Bare syndrome

* Patients must have any B-cell lymphoma, or chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), Gray-zone lymphoma, nodular lymphocyte-predominant Hodgkin lymphoma, or classical Hodgkin lymphoma with any cluster of differentiation 19 (CD19) or cluster of differentiation 20 (CD20) expression on Reed-Sternberg cells. Lower grade lymphomas or CLL transformed to diffuse large B-cell lymphoma (DLBCL) are potentially eligible as is primary mediastinal B-cell lymphoma and all other subtypes of DLBCL. Burkitt and mantle cell lymphoma are potentially eligible.
* For classical Hodgkin lymphoma only, a biopsy from any time from any institution that shows any CD19 or CD20 expression on Reed-Sternberg cells is adequate for eligibility. CD19 or CD20 expression on the Reed-Sternberg cells that is weak or only present on some Reed-Sternberg cells by immunohistochemistry is compatible with protocol eligibility.
* For all lymphoma types except for classical Hodgkin lymphoma, either CD19 or CD20 expression must be uniform. Uniform CD19 or CD20 expression is defined as no obvious lymphoma population lacking antigen expression is present. Antigen expression can be assessed by either immunohistochemistry or flow cytometry.
* Only when insufficient biopsy material is available to allow CD19 and CD20 expression assessment at the National Institutes of Health (NIH), CD19 and/or CD20 staining performed at another institution can be used
* DLBCL patients must have received at least two prior chemotherapy-containing regimens at least one of which must have contained doxorubicin and a monoclonal antibody. Follicular lymphoma patients must have received at least 2 prior regimens including at least 1 regimen with chemotherapy. All other B-cell lymphoma and leukemia patients must have had at least 1 prior chemotherapy-containing regimen. All patients with CLL or small lymphocytic lymphoma must have had prior treatment with ibrutinib or another signal transduction inhibitor and venetoclax.
* Hodgkin lymphoma patients must have:

  * had at least 3 prior lines of therapy.
  * had at least 1 prior cytotoxic chemotherapy-containing regimen.
  * had prior exposure to brentuximab vedotin.
  * had undergone autologous stem cell transplant or been transplant ineligible or refused autologous transplantation
* Eligibility will be expanded to include CD19 and CD20-negative classical Hodgkin lymphoma if any 2 patients with classical Hodgkin lymphoma and CD19/CD20 expression on Reed-Sternberg (RS) cells have durations of response 6 months or greater (responses could be partial responses (PRs) or complete responses (CRs) or a CR of 3 months or greater.
* All patients must have measurable malignancy as defined by at least one of the criteria below.
* Lymphoma or leukemia masses that are measurable (minimum 1.5 cm in largest diameter) by computed tomography (CT) scan is required for all diagnoses except CLL. All masses must be less than or equal to 10.0 cm in the largest diameter.
* For a lymphoma mass to count as measurable malignancy, it must have abnormally increased metabolic activity when assessed by positron emission tomography (PET) scan. CLL masses do not need to have increased activity on positron emission tomography (PET) scan.
* For CLL and lymphoma with only bone marrow involvement no mass is necessary, but if a mass is not present, bone marrow malignancy must be detectable by flow cytometry in lymphoma and CLL. Note that leukemia cells must make up 1% or less of peripheral blood lymphocytes in CLL patients for these patients to be eligible.

OTHER INCLUSION CRITERIA:

* Greater than or equal to 18 years of age.
* Able to understand and sign the Informed Consent Document.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-1
* Room air oxygen saturation of 92% or greater
* Patients of both sexes must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the protocol treatment.
* A patient with a negative blood polymerase chain reaction (PCR) test for hepatitis B deoxyribonucleic acid (DNA) test can be enrolled. If hepatitis B DNA (PCR) testing is not available, patients with a negative hepatitis B surface antigen and negative hepatitis B core antibody can be enrolled.
* Patients must be tested for the presence of Hepatitis C antigen by PCR and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative in order to be eligible. Only if Hepatitis C PCR testing is not available in a timely manner, patients who are Hepatitis C antibody-negative can be enrolled.
* Absolute neutrophil count greater than or equal to 1000/mm^3 without the support of filgrastim or other growth factors.
* Platelet count greater than or equal to 50,000/mm^3 without transfusion support
* Hemoglobin greater than 8.0 g/dl.
* For CLL only, less than or equal to 1% malignant cells in the peripheral blood lymphocytes must be documented by flow cytometry of blood within 2 weeks of protocol enrollment.
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* Serum creatinine less than or equal to 1.5 mg/dl.
* Total bilirubin less than or equal to 2.0 mg/dl.
* Normal cardiac ejection fraction (greater than or equal to 50% by echocardiography) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 4 weeks of treatment start.
* Patients must not take corticosteroids including prednisone, dexamethasone or any other corticosteroid for 14 days before apheresis and chimeric antigen receptors (CAR) T-cell infusion. Patients must also not take corticosteroids at doses higher than 5 mg/day of prednisone or equivalent at any time after the CAR T cell infusion.
* Patients must be able to understand and be willing to sign a written informed consent.
* Patients who have either been previously treated on protocols of genetically-modified T cells on a clinical trial at the National Cancer Institute (NCI) or received T cells modified with the murine stem cell virus-based splice-gag (MSGV) or murine stem cell virus-based splice-gag 1 (MSGV1) gamma-retroviral vectors at any institution are potentially eligible under these conditions:

  * At least 3 months have elapsed since the last genetically-modified T-cell therapy that the patient received, and there is no evidence of replication-competent retroviruses (evidence must be provided from prior protocol Principal Investigator), and persisting genetically-modified T cells are either not detectable in the patient's blood or detectable at levels less than or equal to 0.2% of blood T cells as measured by flow cytometry using the Kip-1 antibody in the flow cytometry lab of the NCI Laboratory of Pathology (Maryalice Stetler-Stevenson's lab).

EXCLUSION CRITERIA:

* Patients that require urgent therapy due to tumor mass effects or spinal cord compression.
* Patients must not have received any anti-CD20 or anti-CD19 antibody products in the past 30 days prior to CAR T-cell infusion.
* Any history of receiving programmed death 1 (PD-1) or programmed death ligand 1 (PD-L1) inhibitors
* Patients that have active hemolytic anemia.
* Human immunodeficiency virus (HIV)-positive patients are excluded because HIV causes complicated immune deficiency and study treatment can pose more risks for these patients.
* Patients with second malignancies in addition to their B-cell malignancy are not eligible if the second malignancy has required treatment (including maintenance therapy) within the past 3 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.

Pregnant women are excluded from this study because study therapy can cause fetal harm. Because there is potential risk for adverse events in nursing infants secondary to treatment of the mother with study therapy, breastfeeding should be discontinued if the mother is treated with study drugs.

* Active uncontrolled systemic infections (defined as infections causing fevers and infections requiring intravenous antibiotics when intravenous antibiotics have been administered for less than 72 hours), active coagulation disorders or other major uncontrolled medical illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary or immune system, history of myocardial infarction, history of ventricular tachycardia or ventricular fibrillation, active cardiac arrhythmias (active atrial fibrillation is not allowed, resolved atrial fibrillation not requiring current treatment is allowed (anticoagulants count as current treatment)), active obstructive or restrictive pulmonary disease, active autoimmune diseases such as rheumatoid arthritis.
* Hospitalization within the 7 days prior to enrollment.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Prior allogeneic stem cell transplant
* Systemic lymphoma treatment of any type and corticosteroid steroid therapy of any dose greater than 5 mg/day or more of prednisone or equivalent is not allowed within 14 days prior to the required leukapheresis, or the initiation of the conditioning chemotherapy regimen. Corticosteroid creams, ointments, and eye drops are allowed.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Patients on systemic anticoagulant therapy except aspirin.
* Active central nervous system metastases or cerebrospinal fluid malignancy. Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Any current neurologic disorders except migraine headaches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Human data will be shared as follows: Coded, linked data in a National Institutes of Health-funded or approved repository. Coded, linked data in the Biomedical Translational Research Information System (BTRIS). And coded, linked or identified data with approved outside collaborators under appropriate agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared before publication and at the time of publication or shortly thereafter indefinitely.
Access Criteria: Data will be shared through ClinicalTrials.gov, BTRIS, approved outside collaborators under appropriate individual agreements, and publication and/or public presentations.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0008.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Principal investigator stopped study due to instability of chimeric antigen receptor gene. | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled on group 2 because the study was stopped. The chimeric antigen receptor (CAR) gene used in this study is prone to recombination events and is therefore not stable.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.95 (12.52) |  | 54.95 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Administered T Cells Expressing a Novel Fully- Human Anti-cluster of Differentiation 19 (CD19) and Anti-cluster of Differentiation 20 (CD20) Chimeric Antigen Receptors (CAR) Who Experienced a Dose-limiting Toxicity (DLT)
Description: A DLT are defined as toxicities assessed by the Common Terminology Criteria for Adverse Events v5.0 that are possibly, probably, or definitely attributable to protocol interventions and occurring between the first protocol treatment through 28 days after the CAR T-cell infusion.
Time Frame: First protocol treatment through 28 days after the CAR T-cell infusion.
Population: 1/2 participants were evaluable on group 1 and no participants were enrolled on group 2. The study was terminated. No participants experienced a DLT probably or definitely attributable to interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
Number analyzed (Participants) | 1 | 0
Participants
  Peripheral Motor Neuropathy Possibly Related | 1 | 0
  Guillain-Barre Syndrome Possibly Related | 1 | 0

2. Secondary Outcome: Percentage of Peak Blood Chimeric Antigen Receptors (CAR) T Cells
Description: We measured CAR T-cell persistence by detecting the CAR gene in peripheral blood mononuclear cells (PBMC) by polymerase chain reaction (PCR).
Time Frame: 119 days after CAR T-cell infusion
Population: 1/2 participants were treated on group 1 and no participants were enrolled on group 2. The study was terminated.
Measure: Number; unit: percentage of PBMC
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
Number analyzed (Participants) | 1 | 0
percentage of PBMC | 10.5 |

3. Secondary Outcome: Percentage of Peripheral Blood Mononuclear Cells (PBMC) of Chimeric Antigen Receptors (CAR) T Cells
Description: Peak blood levels of Chimeric Antigen Receptors (CAR) T cells were measured by exact Wilcoxon rank sum test.
Time Frame: pretreatment and multiple days from day 1 to day 173 after infusion.
Population: 1/2 participants were treated on group 1 and no participants were enrolled on group 2. The study was terminated.
Measure: Number; unit: percentage of PBMC
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
Number analyzed (Participants) | 1 | 0
percentage of PBMC | 10.47 |

4. Secondary Outcome: Number of Participants With Clinical Response
Description: Response for lymphoma was assessed by the Revised Response Criteria for Malignant Lymphoma and The Lugano Classification. Complete Remission (CR) is complete disappearance of all detectable clinical evidence of disease. Partial Remission (PR) is ≥ 50% decrease in nodes or masses. Progressive Disease (PD) is Response ≥ 50% increase in a single node. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor PD. For participants with Chronic Lymphocytic Leukemia (CLL),response was assessed by the International Workshop on CLL. CR is no lymph nodes ≥ 1.5 cm on physical exam or relevant computed tomography. PR is a ≥ 50% decrease in peripheral B lymphocyte count from pre-treatment value. PD is a ≥ 50% increase in the greatest diameter of any lymph node that was enlarged pretreatment. And SD are participants who do not fulfill the criteria for CR, PR or PD.
Time Frame: Approximately 1 year 5 months
Population: 1/2 participants were evaluable on group 1 and no participants were enrolled on group 2 because the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
Number analyzed (Participants) | 1 | 0
Participants
  Complete Remission | 0 |
  Partial Remission | 1 |
  Progressive Disease | 0 |
  Stable Disease | 0 |

5. Secondary Outcome: Last Time-Point at Which Chimeric Antigen Receptors (CAR) T Cells Were Detected in the Blood
Description: Chimeric Antigen Receptors (CAR) T cell persistence was measured in the blood by quantitative polymerase chain reaction (PCR). CAR T cells that are detected in the participant's blood that persist for a significant length of time is a positive finding.
Time Frame: 119 days after CAR T-cell infusion
Population: 1/2 participants were treated on group 1 and no participants were enrolled on group 2. The study was terminated.
Measure: Number; unit: Days
Groups:
- 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation: All patients will be receiving escalating dose of Anti-cluster of differentiation 19 (CD19) and anti-cluster of differentiation 20 (CD20) CAR T cells/kg + conditioning chemotherapy
  Anti-cluster of differentiation 19 (CD19)-Chimeric Antigen Receptors (CAR) and Anti-cluster of differentiation 20 (CD20)-CAR T cells: Dose-escalation trial starting dose: 0.66 x10^6 CAR+ T cells/kg (weight-based dosing one time) (up to a maximum dose of 10x10^6 CAR+ T cells/kg based on cohort) infuse on day 0
  Cyclophosphamide: 500 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3
  Fludarabine: 30 mg/m^2 intravenous (IV) infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
Number analyzed (Participants) | 1 | 0
Days | 119 |

6. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 7 months and 18 days.
Population: 1/2 participants were treated on group 1 and no participants were enrolled on group 2. The study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

7. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD) of Chimeric Antigen Receptors (CAR) T Cells
Description: The maximum tolerated dose is the dose at which a maximum of 1 of 6 participants has a dose-limiting toxicity (DLT). A DLT are defined as toxicities that are possibly, probably, or definitely attributable to protocol interventions and occurring between the first protocol treatment through 28 days after the CAR T-cell infusion.
Time Frame: First protocol treatment through 28 days after the CAR T-cell infusion.
Measure: Number; unit: T cells
Groups:
- All Participants: All participants treated on 1/Conditioning chemotherapy plus Chimeric Antigen Receptors (CAR) T-cells dose escalation and 2/Conditioning chemotherapy plus Chimeric Antigen Receptors (CAR) T-cells expansion phase.
Arm/Group | All Participants
Number analyzed (Participants) | 1
T cells | NA — The MTD was not found because 1/2 participants were treated on group 1 and no participants were enrolled on group 2. The study was terminated.

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 7 months and 18 days.
Description: No participants were enrolled on group 2 because the study was stopped. The chimeric antigen receptor (CAR) gene used in this study is prone to recombination events and is therefore not stable. And 1/2 participants were treated on group 1.
Arm/Group | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation (N=1) | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase (N=0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — cervical lymph node biopsy showed squamous cell carcinoma
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Dose Escalation (N=1) | 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptors (CAR) T-cells Expansion Phase (N=0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (13) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (6) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (16) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (6) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT04160195/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT04160195/ICF_001.pdf